CLINICAL TRIAL: NCT02757482
Title: Effects of Patient Training About the Safety of Warfarin Therapy on the Patients' Warfarin Knowledge Level and International Normalized Ratio Control (INR)
Brief Title: Patient Training About the Safety of Warfarin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Tülay SAĞKAL MİDİLLİ, Asistant professor, Asistant Professor, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CBU-2015-02
Record Dates: First submitted 2016-04-24; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Warfarin Knowledge Level; International Normalized Ratio Control; Patient Training
Keywords: Patient training; Warfarin; International Normalized Ratio; Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Patient training
  Interventions: Other: training
- control (No Intervention): no patient training

INTERVENTIONS:
Other: training
  Arms: intervention

SUMMARY:
The purpose of this study is to examine the effects of patient training about the safety of warfarin therapy on related knowledge levels and on International Normalized Ratio (INR) control.

DETAILED DESCRIPTION:
Although warfarin is widely used in the treatment and prophylaxis of thromboembolic diseases, it is an oral anticoagulant with serious adverse effects. Therefore, the patient must be informed about its safe use.

A patient's level of knowledge concerning the drug plays a key role in the effective and safe use of warfarin. In the Joint Commission International (JCI) National Patient Safety Goal (NPSG) guideline for 2014 education on treatment for patients taking oral anticoagulants was recognized as a vital factor. Previous studies have reported that a positive relationship between patients' anticoagulant knowledge levels and the INR number in the therapeutic range.

For this reason there is a need for effective education programs to increase patients' knowledge concerning warfarin and to keep it up to date. Education and information services provided to patients using anticoagulants will reduce the costs of treatment by reducing risks such as thromboembolism and bleeding. When planning education, individual characteristics and needs must be kept in mind, and group education in addition to individual sessions and the use of written and visual material will increase the effectiveness of the education.

ELIGIBILITY:
Inclusion Criteria:

* Using warfarin for at least two months,
* Between 18 and 65 years old,
* Were literate,
* Not have a structured education about warfarin

Exclusion Criteria:

* Have structured education about warfarin,
* Have a seeing or hearing disability,
* Have a cognitive or sensory disorder,
* Have a disability affecting oral communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Warfarin Knowledge Level Measurement | 2 months
  Warfarin knowledge level was measured by The Warfarin Knowledge Assessment Form. This form consisted of 30 questions. These questions covered basic information for drug treatment such as the drug dose, the duration of drug use, adverse effects of the drug, drug-drug and drug-food interaction, drug use in pregnancy, dental care and treatment, laboratory monitoring, exercise and diet. Each correct answer scored 1, and each wrong answer or a 'don't know' response scored 0. The last two questions in the last section on drug use related to pregnancy and nursing a child, and so these were answered only by women. Patients' raw information scores were between 0 and 30. Those scoring 0-15 were accepted as having a low level of information, those scoring 16-21 a moderate level, and those scoring 22-30 a high level of information.

SECONDARY OUTCOMES:
International Normalized Ratio Measurements | 6 months
  The last three INR measurement values for the two patient groups were taken from the hospital records and recorded, together with the INR values for the day of the first interview. The warfarin knowledge evaluation form was applied again to the patients of each group in the first and second months, and the INR values for those dates were obtained from hospital records.

CONTACTS AND LOCATIONS:
Overall Officials: TULAY SAGKAL MIDILLI, Phd, RN, Study Director — Assistant professor
Locations (1):
- CELAL BAYAR UNIVERSITY Ö.Y.P. (Teaching Staff Training Program) OFFICE, Manisa, Muradiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided